CLINICAL TRIAL: NCT05546307
Title: Randomized, Single-blind Study Evaluating the Interest of Prior Relaxation on the Quality of the Recordings of the SomatoSensory Evoked Potentials
Brief Title: Interest of Prior Relaxation on the Recordings of the SomatoSensory Evoked Potentials
Acronym: RELAXPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2019_843_0079
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Relaxation; Somatosensory Evoked Potentials; Patient Experience
Keywords: Relaxation; Somatosensory Evoked Potentials; Patient experience

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- one relaxation session before the examination (Experimental)
  Interventions: Other: SSEP; Other: relaxation session
- No relaxation session before the examination (Active Comparator)
  Interventions: Other: SSEP

INTERVENTIONS:
Other: SSEP — Every patient presenting for a SSEP will be offered to participate to the study. If accepted, a randomization will determine whether the examination will be preceded by a relaxation session (Relax Group) or not (control group)
Other: relaxation session — The relaxation session will be performed by one of the 5 nurses trained in relaxation
  Arms: one relaxation session before the examination

SUMMARY:
Many factors influence the quality and duration of SomatoSensory Evoked potentials (SSEP). Some are related to the technique : type of electrodes, intensity of stimulation, stimulation site ; others are related to the patient : poor state of relaxation of the patient generating muscle artefacts; hypersensitivity of the patient to electrical stimuli making the examination unpleasant; examination time considered too long. However, the patient's relaxed state is essential to the quality of the signal . Thus the duration of an examination is very variable : between 30 and 75 minutes for the upper limbs.... For several months, the investigators provide relaxation to some patients just before the examination. Results seem to be positive. The investigators aim to study the effect of relaxation session on the quality of the SSEP recordings. Fifteen-minutes relaxation session will be provided by a nurse trained to the relaxation.

The investigators will compare two groups : one group with one relaxation session before the examination and one group without relaxation session before the examination.

The investigators chose to study the influence of relaxation session on (i) the artifacts rejection rate by the machine for the recordings of SSEP by stimulation of the median nerve to the upper limbs (ii) the duration of the examination (iii) the patient experience

ELIGIBILITY:
Inclusion Criteria:

* Any patient addressed for a study of the somatosensory evoked potentials in upper limbs
* Patients between 18 to 70 years old.
* Patients able to understand the instructions of the relaxation session and the examination.
* Patient providing informed consent exclusion criteria

Exclusion Criteria:

* No availability of a technician trained in relaxation
* Patient's refusal to participate in the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Variation of average rate of automatized artifacts rejection between both groups | 19 months
  Average rate of automatized artifacts rejection during 2 sessions of 1000 stimulations on the first stimulated limb to obtain the N13 wave

CONTACTS AND LOCATIONS:
Locations (1):
- Amiens University Hospital, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No